CLINICAL TRIAL: NCT06486363
Title: Comparison of the Antiplatelet Efficacy of Aspirin Combined With Clopidogrel and Aspirin Combined With Half-dose Ticagrelor in Patients With Unruptured Intracranial Aneurysms With Normal CYP2C19 Metabolizer Phenotype
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Shijie Na, Deputy chief physician of Neurosurgery, Principal Investigator, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-536-02
Record Dates: First submitted 2024-06-19; First posted 2024-07-03 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Intracranial Aneurysms; Antiplatelet Drugs
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Clopidogrel

STUDY DESIGN:
Intervention Model Description: To compare the antiplatelet efficacy of aspirin combined with clopidogrel and aspirin combined with half-dose ticagrelor in in patients with unruptured intracranial aneurysms with normal CYP2C19 metabolizer phenotype
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin combined with clopidogrel (Active Comparator): Participants in this group shall take Aspirin (100 mg/day) + clopidogrel (75 mg/day) for at least 5 days before receiving stent-assisted coil embolization, and take same medication for 6 months after endovascular treatment
  Interventions: Drug: Aspirin combined with clopidogrel
- Aspirin combined with half-dose ticagrelor (Experimental): Participants in this group shall take Aspirin (100 mg/day) + half dose of ticagrelor (45 mg, 12 hours/time), at least for 3 days before receiving stent-assisted coil embolization, and take same medication for 6 months after endovascular treatment.
  Interventions: Drug: Aspirin combined with half-dose ticagrelor

INTERVENTIONS:
Drug: Aspirin combined with clopidogrel — Participants in this group shall take Aspirin (100 mg/day) + clopidogrel (75 mg/day) for at least 5 days before receiving stent-assisted coil embolization, and take same medication for 6 months after endovascular treatment
  Arms: Aspirin combined with clopidogrel
Drug: Aspirin combined with half-dose ticagrelor — Participants in this group shall take Aspirin (100 mg/day) + half dose of ticagrelor (45 mg, 12 hours/time), at least for 3 days before receiving stent-assisted coil embolization, and take same medication for 6 months after endovascular treatment
  Arms: Aspirin combined with half-dose ticagrelor

SUMMARY:
The goal of this clinical trial is to compare the antiplatelet efficacy of aspirin combined with clopidogrel and aspirin combined with half-dose ticagrelor in in patients with unruptured intracranial aneurysms with normal CYP2C19 metabolizer phenotype. The main questions it aims to answer are:

If aspirin combined with half-dose ticagrelor is comparable to or better than aspirin combined with clopidogrel? What medical problems do participants have when taking aspirin combined with half-dose ticagrelor? Researchers will compare aspirin combined with half-dose ticagrelor to aspirin combined with clopidogrel to see if aspirin combined with half-dose ticagrelor works to treat patients with unruptured intracranial aneurysms received endovascular treatment.

Participants will:

Take aspirin combined with half-dose ticagrelor or aspirin combined with clopidogrel every day for 6 months Visit the clinic 1 month and 6 months for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unruptured intracranial aneurysms who are scheduled for stent-assisted embolization;
2. mRS score less than or equal to 2 on admission;
3. Normal CYP2C19 metabolizer genotype;
4. Age 20 or above, 70 or below, regardless of gender;
5. The subject or the entrusted family member voluntarily signed the informed consent for this trial

Exclusion Criteria:

1. Use of drugs that affect coagulation function or significant abnormalities in platelet/coagulation function before admission;
2. Previous history of cardiovascular and cerebrovascular disease;
3. Complications of major organ dysfunction, chronic inflammatory diseases or malignant tumors at admission;
4. Known allergy or contraindication to heparin, aspirin, clopidogrel, or ticagrelor;
5. Patients with any severe or active pathological bleeding;
6. Pregnant and lactating female;
7. Those deemed unsuitable to participate in this trial by the responsible physician

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of cerebral stroke | The entire experimental process after endovascular treatment
  Incidence rate of cerebral stroke, including ischemic stroke and hemorrhagic stroke
Modified Rankin Scale | 6 months after endovascular surgery
  Modified Rankin Scale ( The scale runs from 0 to 6, 0 means perfect health and 6 means death)
Mini-mental state examination | 6 months after endovascular surgery
  The MMSE examination includes time and place orientation, registration, attention and calculation, recall, language, repitition, complex commands. Score excess 24 or more indicates a normal cognition, 19-23 points indicates mild cognitive impairment, score of 10-18 points indicates moderate cognitive impairment and score below 9 points indicates severe cognitive impairment

SECONDARY OUTCOMES:
Platelet inhibition rate/platelet aggregation rate | 1 day before endovascular surgery/3 days after endovascular surgery/3 and 6 months after endovascular surgery
  Platelet inhibition rate/platelet aggregation rate

CONTACTS AND LOCATIONS:
Overall Officials: Shijie Na, Doctor, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing university

IPD SHARING:
Plan to Share IPD: No